CLINICAL TRIAL: NCT06043713
Title: Phase I Study of Autologous CD8+ and CD4+ Transgenic T Cells Expressing High Affinity KRASG12V Mutation-Specific T Cell Receptors in Participants With Metastatic Solid Tumors With KRAS G12V Mutations
Brief Title: Autologous CD8+ and CD4+ Transgenic T Cells Expressing High Affinity KRASG12V Mutation-Specific T Cell Receptors (FH-A11KRASG12V-TCR) in Treating Patients With Metastatic Solid Tumor Cancers With KRAS G12V Mutations
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Affini-T Therapeutics, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1123135; NCI-2023-06287 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20048 (Other: Fred Hutch/University of Washington Cancer Consortium); 2P50CA228944 (NIH)
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Bendamustine Hydrochloride; Biopsy; Specimen Handling; Cyclophosphamide; fludarabine; Leukapheresis; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (FHA11KRASG12V-TCR) (Experimental): Patients undergo leukapheresis prior to treatment and receive lymphodepletion chemotherapy with either cyclophosphamide IV and fludarabine IV on days -6, -5, and -4, or bendamustine IV on days -4 and -3 at the discretion of the treating clinician and/or PI. Patients then receive FHA11KRASG12V-TCR IV on day 0. Patients may receive an additional FHA11KRASG12V-TCR IV infusion as soon as 28 days or up to 1 year after the first infusion. Patients undergo ECHO or MUGA during screening. Patients also undergo CT, PET or MRI as well as blood sample collection and a tissue biopsy at baseline and throughout the trial.
  Interventions: Drug: Bendamustine; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography; Drug: Fludarabine; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Biological: T-cell Receptor-engineered T-cells

INTERVENTIONS:
Drug: Bendamustine — Receive IV
  Other Names: SDX-105
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Cyclophosphamide — Receive IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Fludarabine — Receive IV
  Other Names: Fluradosa
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning; RNV Scan
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: T-cell Receptor-engineered T-cells — Receive FHA11KRASG12V-TCR IV
  Other Names: T-cell Receptor-engineered T Cells; T-cell Receptor-engineered T-lymphocytes; TCR T Cells; TCR T-cells; TCR-engineered T-cells; TCR-modified T Cells; FH-A11KRASG12V-TCR; AFNT-111

SUMMARY:
This phase I trial studies the side effects and best dose of autologous CD8+ and CD4+ transgenic T cells expressing high affinity KRASG12V mutation-specific T cell receptors (FH-A11KRASG12V-TCR) and to see how well they work in treating patients with solid tumor cancers that has spread from where it first started (primary site) to other places in the body (metastatic). T cells are infection fighting blood cells that can kill tumor cells. The T cells given in this study will come from the patient and will have a new gene put in them that makes them able to recognize KRAS G12V, a protein on the surface of tumor cells. These KRAS G12V-specific T cells may help the body's immune system identify and kill KRAS G12V solid cancer tumor cells.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of FHA11KRASG12V-TCR.

Patients undergo leukapheresis prior to treatment and receive lymphodepletion chemotherapy with either cyclophosphamide intravenously (IV) and fludarabine IV on days -6, -5, and -4, or bendamustine IV on days -4 and -3 at the discretion of the treating clinician and/or principal investigator (PI). Patients then receive FHA11KRASG12V-TCR IV on day 0. Patients may receive an additional FHA11KRASG12V-TCR IV infusion as soon as 28 days or up to 1 year after the first infusion. Patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening. Patients also undergo computed tomography (CT), positron emission tomography (PET) or magnetic resonance imaging (MRI) as well as blood sample collection and a tissue biopsy at baseline and throughout the trial.

After completion of study treatment, patients are followed up on day 56, 112, 168, 224, 280 and day 365, then long-term for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* LEUKAPHERESIS: Diagnosis of metastatic solid tumor
* LEUKAPHERESIS: Tissue confirmation of solid tumor. Confirmation of diagnosis must be or have been performed by internal pathology review of archival biopsy material or other pathologic material at Fred Hutch/University of Washington Cancer Consortium (UWMC)
* LEUKAPHERESIS: HLA-A*11:01 confirmed through HLA typing at a clinically accredited laboratory
* LEUKAPHERESIS: Previously documented KRASG12V mutation in tumor or plasma cell-free deoxyribonucleic acid (cfDNA) specimens by polymerase chain reaction (PCR) or next-generation sequencing (NGS) test
* LEUKAPHERESIS: Measurable disease by RECIST 1.1 criteria: Participants must have measurable disease, defined as at least one target lesion that can be measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm, unless lymph node in which case short axis must be ≥ 15 mm. Baseline imaging (for example, diagnostic CT chest/abdomen/pelvis and imaging of the affected extremity as appropriate), brain imaging (MRI or CT scan) if clinically indicated, must be obtained within 8 weeks of the first planned T cell infusion. MRI can be substituted for CT in participants unable to have CT contrast
* LEUKAPHERESIS: Participants must be willing to undergo tumor biopsy for research purposes if safe and feasible at baseline (prior to first T cell infusion), 2-3 weeks after the first T cell infusion, and approximately 2 weeks +/- 1 week after the 2nd infusion (if applicable), if safe and feasible (these time windows may vary due to manufacturing or clinical reasons). Should there be no tumor tissue that is accessible for biopsy, subjects will still be considered for participation, at the discretion of the investigator. Similarly, should an investigator determine that a biopsy cannot be performed safely for clinical reasons, biopsies may be cancelled or rescheduled. Patients can also refuse biopsies at any time after enrollment
* LEUKAPHERESIS: Participants must be at least two weeks or five half-lives (for small molecules) from last systemic treatment: At least 2 weeks must have passed since any: immunotherapy (for example, T-cell infusions, immunomodulatory agents, interleukins, vaccines), or chemotherapy cancer treatment. At least five half-lives must have passed from treatment with small molecules or other investigational agents. There is no washout period for radiation, so long as radiated lesion is not the lesion being evaluated for RECIST measurements on the protocol. Bisphosphonates and denosumab are permitted
* LEUKAPHERESIS: Participants must have progressed on or be intolerant to at least one lines of prior therapy including any targeted therapies indicated for subjects with each of the tumor types eligible to enroll, as applicable
* LEUKAPHERESIS: Patients with solid tumors harboring targetable molecular alterations including but not limited to EGFR mutations, ALK, ROS, NTRK fusions, microsatellite instability (MSI)-high, tumor mutational burden (TMB) high, BRAF v600 mutations, HER2 amplifications, must have been treated or refused treatment with applicable targeted therapies, as applicable
* LEUKAPHERESIS: Fertile male and female participants must be willing to use an effective contraceptive method before, during, and for at least 4 months after the last A11KRASG12V-TCR infusion
* LEUKAPHERESIS: 18 years or older at the time of enrollment
* LEUKAPHERESIS: Capable of understanding and providing a written informed consent
* LEUKAPHERESIS: Eastern Cooperative Oncology Group (ECOG) performance status of =< 1

  * No uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage more than once every 28 days
* LEUKAPHERESIS: No uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage more than once every 28 days
* LEUKAPHERESIS: Renal: Creatinine clearance >= 50 ml/min by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) or 24-hour urine clearance
* LEUKAPHERESIS: Hepatic: Total bilirubin < 2.0 mg/dL
* LEUKAPHERESIS: Hepatic: Aspartate transferase (AST) and alanine transaminase (ALT) < 5x upper limit of normal (ULN)
* LEUKAPHERESIS: Hepatic: Participants with suspected Gilbert syndrome may be included if total bilirubin (Bili) > 3 mg/dL but no other evidence of hepatic dysfunction
* LEUKAPHERESIS: Cardiac: Participants 60 years of age or older are required to have left ventricular ejection fraction (LVEF) evaluation performed within 60 days prior to enrollment. LVEF may be established with echocardiogram or MUGA scan, and LVEF must be >= 35%. Cardiac evaluation for other participants is at the discretion of the treating physician
* LEUKAPHERESIS: Hematologic: Absolute neutrophil count (ANC) >= 1000 cells/ mm^3
* LEUKAPHERESIS: Nutrition: Albumin >= 3 g/dL
* START OF TREATMENT: Measurable disease by RECIST 1.1 criteria: Participants must have measurable disease, defined as at least one target lesion that can be measured in at least one dimension (longest diameter to be recorded) as >= 10 mm, unless lymph node in which case short axis must be >= 15 mm. Baseline imaging (for example, diagnostic CT chest/abdomen/pelvis and imaging of the affected extremity as appropriate), brain imaging (MRI or CT scan) must be obtained within 8 weeks of the first planned T cell infusion. MRI can be substituted for CT in participants unable to have CT contrast
* START OF TREATMENT: Participants must be willing to undergo tumor biopsy for research purposes if safe and feasible at baseline (prior to first T cell infusion), 2-3 weeks after the first T cell infusion, and approximately 2 weeks +/- 1 week after the 2nd infusion (if applicable), if safe and feasible (these windows may vary due to manufacturing or clinical reasons). Should there be no tumor tissue that is accessible for biopsy, subjects will still be considered for participation, at discretion of the investigator. Similarly, should an investigator determine that a biopsy cannot be performed safely for clinical reasons, biopsies may be cancelled or rescheduled
* START OF TREATMENT: Participants must be at least two weeks from last systemic treatment: At least 2 weeks must have passed since any: immunotherapy (for example, T-cell infusions, immunomodulatory agents, interleukins, vaccines), or chemotherapy cancer treatment. At least five half-lives must have passed from treatment with small molecules or other investigational agents. There is no washout period for radiation, so long as radiated lesion is not the lesion being evaluated for RECIST measurements on the protocol. Bisphosphonates and denosumab are permitted
* START OF TREATMENT: ECOG performance status of =< 1
* START OF TREATMENT: Renal: Creatinine clearance >= 50 ml/min by CKD-EPI or 24-hour urine clearance

  * Exceptions may be at the discretion of the PI to allow participants with organ function affected by their organ-specific tumor involvement
* START OF TREATMENT: Hepatic: Total bilirubin < 2.0 mg/dL

  * Exceptions may be at the discretion of the PI to allow participants with organ function affected by their organ-specific tumor involvement
* START OF TREATMENT: AST and ALT < 5x upper limit of normal (ULN)
* START OF TREATMENT: Participants with suspected Gilbert syndrome may be included if total Bili > 3 mg/dl but no other evidence of hepatic dysfunction
* START OF TREATMENT: Pulmonary: =< grade 1 dyspnea and oxygen saturation of arterial blood (SaO2) >= 92% on ambient air. If pulmonary function tests (PFTs) are performed based on the clinical judgement of the treating physician, participants with forced expiratory volume in the first second (FEVI) >= 50% of predicted and diffusing capacity of the lungs for carbon monoxide (DLCO) (corrected) >= 40% of predicted will be eligible

  * Exceptions may be at the discretion of the PI to allow participants with organ function affected by their organ-specific tumor involvement
* START OF TREATMENT: Hematologic: ANC >= 1000 cells/ mm^3

  * Exceptions may be at the discretion of the PI to allow participants with organ function affected by their organ-specific tumor involvement
* START OF TREATMENT: Nutrition: Albumin >= 3 g/dL

  * Exceptions may be at the discretion of the PI to allow participants with organ function affected by their organ-specific tumor involvement
* START OF TREATMENT: Participants with a history of chronic obstructive pulmonary disease (COPD), emphysema, or greater than 30 pack year smoking history should undergo PFTs and meet the following criteria:

  * FEVI >= 50% of predicted and DLCO (corrected) >= 40% of predicted will be eligible

Exclusion Criteria:

* LEUKAPHERESIS: Prior solid organ transplant or allogeneic hematopoietic stem cell transplant: Kidney transplant participants will be considered on a case-by-case basis requiring discussion with PI. If the participant has had a kidney transplant, participant must have dialysis access, dialysis plan, supportive nephrologist, willingness to stop transplant immunosuppression, and express understanding that rejection is possible outcome. Dialysis or costs related to transplant kidney will not be supported by the study. Participants having had any other solid organ transplants will be excluded, as will those with any history of allogeneic hematopoietic stem cell transplant
* START OF TREATMENT: Pregnancy, breastfeeding, or expecting to conceive or father children for the duration of the trial through 4 months after last T-cell infusion. Participants of childbearing potential must have a negative serum pregnancy test within the 2 weeks (14 days) preceding T cell infusion. Childbearing potential is defined as women who have not been surgically sterilized and who are not post-menopausal (free of menses for at least 1 year)
* START OF TREATMENT: Active autoimmune disease: Participants with active autoimmune disease requiring immunosuppressive therapy are excluded. Case by case exemptions are possible with approval by PI
* START OF TREATMENT: Corticosteroid therapy at a dose equivalent of > 0.5 mg/kg of prednisone per day. The following treatments are permitted: intranasal, inhaled, topical, or local steroid applications; systemic corticosteroids at physiologic doses equivalent to no more than > 0.5 mg/kg/day prednisone; steroids as premedication for contrast dye allergy
* START OF TREATMENT: Concurrent use of other investigational anti-cancer agents
* START OF TREATMENT: Active uncontrolled infection: Human immunodeficiency virus (HIV) positive participants on highly active antiretroviral therapy (HAART) with a CD4 count > 500 cells/mm^3 are considered controlled, as are individuals with a history of hepatitis C who have successfully completed antiviral therapy with an undetectable viral load, and those with hepatitis B who have hepatitis well controlled on medication
* START OF TREATMENT: Uncontrolled concurrent illness: Participants may not have uncontrolled or concurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* START OF TREATMENT: Untreated brain metastases: Participants with small asymptomatic brain metastases (< 1 cm) or those with brain metastases previously treated and controlled with surgery or radiotherapy will be considered for inclusion at discretion of PI, so long as all other eligibility criteria are met
* START OF TREATMENT: Active treatment for prior immune related adverse event to any immunotherapy: Participants receiving ongoing treatment for prior serious immune-related adverse events are excluded, with exception of hormone supplementation or corticosteroid therapy at equivalent of up to 0.5mg/kg/day prednisone per day, unless otherwise approved by PI
* START OF TREATMENT: Other medical, social, or psychiatric factor that interferes with medical appropriateness and/or ability to comply with study, as determined by the PI
* START OF TREATMENT: Known allergic reactions to any of the components of study treatments
* START OF TREATMENT: Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage more than once every 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Within 1 year after 1st infusion of (autologous CD8+ and CD4+ transgenic T cells expressing high affinity KRASG12V mutation-specific T cell receptors (FH-A11KRASG12V-TCR)
  Safety and tolerability should be evaluated after each infusion. Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0).
Dose-limiting toxicity rates | From the time of lymphodepletion chemotherapy to 28 days after FH-A11KRASG12V-TCR infusion
  Will be assessed by treatment-related grade 3 or higher toxicity and assessed by NCI CTCAE v5.0. The treatment will be considered to have an acceptable safety profile if the observed toxicity rate is consistent with a true rate that does not exceed 35%.
Maximum tolerated dose of FH-A11KRASG12V-TCR | From the time of lymphodepletion chemotherapy to 28 days after FH-A11KRASG12V-TCR infusion
  Will be assessed by NCI CTCAE v5.0.
Recommended phase 2 dose of FH-A11KRASG12V-TCR | Within 1 year after 1st infusion of FH-A11KRASG12V-TCR
  Will be assessed by NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Reproducibly generating FHA11KRASG12V- TCR from autologous participant cells (Feasibility) | Within 1 year after eligibility determination
  Defined as the ability to reproducibly generate and infuse the T cells for eligible participants and a simple estimate of the proportion along with its 95% confidence interval will be used. Standard methods will be used to estimate each of the secondary endpoints.
Overall response rate (ORR) | Within 1 year after 1st infusion of FH-A11KRASG12V-TCR
  Will be assessed by complete (CR) and partial responses (PR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria in treated individuals. Standard methods will be used to estimate each of the secondary endpoints.
Stable disease (SD) | Within 1 year after 1st infusion of FH-A11KRASG12V-TCR
  Will be assessed by RECIST 1.1 criteria in treated individuals. Standard methods will be used to estimate each of the secondary endpoints.
Clinical benefit rate (CBR) | Within 1 year after 1st infusion of FH-A11KRASG12V-TCR
  CBR will be defined as ORR + SD. Will be assessed by RECIST 1.1 criteria in treated individuals. Standard methods will be used to estimate each of the secondary endpoints.
ORR | Within 1 year after 1st infusion of FH-A11KRASG12V-TCR
  Will be assessed by immune RECIST 1.1 criteria in treated individuals. Standard methods will be used to estimate each of the secondary endpoints.
Progression-free survival | From study registration to disease progression or death of any cause), assessed up to 1 year after 1st infusion of FH-A11KRASG12V-TCR
  Will be estimated using the method of Kaplan and Meier, with time zero the time of study registration. Standard methods will be used to estimate each of the secondary endpoints.
Overall survival | From study registration to death of any cause, assessed up to 1 year after 1st infusion of FH-A11KRASG12V-TCR
  Will be estimated using the method of Kaplan and Meier, with time zero the time of study registration. Standard methods will be used to estimate each of the secondary endpoints.
Changes in tumor microenvironment | Within 1 year after 1st infusion of FH-A11KRASG12V-TCR
  Will be assessed including immune cells phenotype and collagen or cancer associated fibroblasts in tumor biopsies. Standard methods will be used to estimate each of the secondary endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Chiorean, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT06043713/ICF_000.pdf